CLINICAL TRIAL: NCT02177643
Title: Effect of Diacerein in the Metabolic Control of Patients With Diabetes Mellitus Type 2 and Secondary Failure to Metformin
Brief Title: Effect of Diacerein in the Metabolic Control of Patients With DM Type 2 and Secondary Failure to Metformin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); ANS Pharma (Industry)
Responsible Party: Principal Investigator, Aleksandra Alves Silva, Study Director - Dr. Mario José Abdalla Saad - National Institute of Science and Technology of Obesity and Diabetes, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07943212.5.2002.0053; CAAE: 07943212.5.2002.0053 (Other: National Committee for Ethics in Research - CEP/CONEP BRAZIL)
Record Dates: First submitted 2014-06-23; First posted 2014-06-27 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes-Related Complications; Diabetes Mellitus, Type 2; Insulin Resistance
Keywords: Diabetes; Diacerein
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus, Type 2; Insulin Resistance; Diabetes Mellitus | interventions — diacerein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diacerein (Active Comparator): Diacerein 50 mg immediate release capsule, once daily for the starting 28 days and Diacerein 50 mg immediate release capsule twice a day for the remains of the study.
  Interventions: Drug: Diacerein
- Placebo (Placebo Comparator): Placebo capsules once a day for the starting 28 days and two times daily for the remainder of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diacerein — Diacerein oral capsules
  Other Names: Artrodar - TRB Pharma
  Arms: Diacerein
Drug: Placebo — Placebo oral capsules
  Arms: Placebo

SUMMARY:
Considering that, Diacerein is on the market for almost 20 years, being used continuously in elderly patients with osteoarthritis without present significant side effects, and considering the anti-hyperglycemic effect and the improvement in the insulin resistance observed in animal models of type 2 diabetes and in a previously study from Mexico. The aim of our study is to investigate the effect of Diacerein, a medication with anti-osteoarthritic properties and moderately analgesic activity, anti-inflammatory and antipyretic, which demonstrates inhibit properties for the synthesis of pro-inflammatory cytokines such as interleukin 1 (IL-1). Administered for 12 weeks and the effect in the glycemic and metabolic control in patients with diabetes mellitus 2 and secondary failure to metformin treatment.

DETAILED DESCRIPTION:
This proof of concept study aims to access the metabolic control in patients with type 2 diabetes mellitus and secondary failure to metformin.

The Study is a Phase II, Multicenter, National, Prospective, Randomized, Double blind, Parallel Groups, Placebo Comparative Trial. UNICAMP (Hospital of Unicamp) is the coordinating center and we have the participation of the State University of Feira de Santana and the Center for Diabetes and Hypertension in Fortaleza.

Study Objectives: To investigate the effect of Diacerein administered for 12 weeks; glycemic and metabolic control in patients with diabetes mellitus 2 and secondary failure to metformin treatment. The Total Number of patients will be approximately 60, 30 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus (DM) type 2 between 6 months to 10 years of disease
* Body mass index between 25 and 35 kg/m2
* Fasting glucose between 120 and 250 mg/dL
* Glycated Hb A1c greater than 7,5 %
* Taking Metformin (dose above 1700 mg/day) with or without other secretagogue.

Exclusion Criteria:

* Subjects with DM1
* Subjects with DM2 using insulin
* Subjects with DM2 with chronic complications that already have clinical consequences
* Subjects with other types of diabetes
* Creatinine serum greater than 1.4 mg/dl (female) and 1.5 mg/dl (male)
* History of heart disease and/or severe concomitant diseases such as liver, coronary artery, renal
* History of severe psychiatric or neurological disorders
* History of alcohol abuse and/or illegal drugs or psychotropic medicines in the past six months
* Hypersensitivity to any component of the of study drug and placebo formulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Fasting Glucose Concentration | Baseline, 12 weeks
Fasting Insulin Concentration | Baseline, 12 weeks
HbA1c - glycated haemoglobin | Baseline, 12 weeks
Inflammatory Activity Profile | Baseline, 12 weeks
  TNFα IL6 IL1β C-Reactive Protein (CRP)
Lipid Panel | Baseline, 12 weeks
Hepatic Function Panel | Baseline, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mario JA Saad, MD PhD, Study Director — National Institute of Science and Technology of Obesity and Diabetes (CNPq)
Locations (3):
- Brazil (3):
  - Centro de Estudos em Diabetes e Hipertensão, Fortaleza, Ceará
  - Universidade Estadual de Feira de Santana, Feira de Santana, Estado de Bahia
  - Universidade Estadual de Campinas, Campinas, São Paulo

REFERENCES:
- [Background] Ramos-Zavala MG, Gonzalez-Ortiz M, Martinez-Abundis E, Robles-Cervantes JA, Gonzalez-Lopez R, Santiago-Hernandez NJ. Effect of diacerein on insulin secretion and metabolic control in drug-naive patients with type 2 diabetes: a randomized clinical trial. Diabetes Care. 2011 Jul;34(7):1591-4. doi: 10.2337/dc11-0357. Epub 2011 May 24. PMID 21610123
- [Background] Tobar N, Oliveira AG, Guadagnini D, Bagarolli RA, Rocha GZ, Araujo TG, Prada PO, Saad MJ. Comment on: Ramos-Zavala et al. Effect of diacerein on insulin secretion and metabolic control in drug-naive patients with type 2 diabetes: a randomized clinical trial. Diabetes Care 2011;34:1591-1594. Diabetes Care. 2012 Feb;35(2):e13; author reply e14. doi: 10.2337/dc11-1856. No abstract available. PMID 22275450
- [Background] Tobar N, Oliveira AG, Guadagnini D, Bagarolli RA, Rocha GZ, Araujo TG, Santos-Silva JC, Zollner RL, Boechat LH, Carvalheira JB, Prada PO, Saad MJ. Diacerhein improves glucose tolerance and insulin sensitivity in mice on a high-fat diet. Endocrinology. 2011 Nov;152(11):4080-93. doi: 10.1210/en.2011-0249. Epub 2011 Sep 6. PMID 21896669
- [Background] Velloso LA, Folli F, Perego L, Saad MJ. The multi-faceted cross-talk between the insulin and angiotensin II signaling systems. Diabetes Metab Res Rev. 2006 Mar-Apr;22(2):98-107. doi: 10.1002/dmrr.611. PMID 16389635